CLINICAL TRIAL: NCT06178679
Title: A Phase 3 Multi-Center, Randomized, Double Masked, Vehicle Controlled Study to Assess the Safety and Efficacy of ST-100 (Vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution in Subjects Diagnosed With Dry Eye Disease (DED)
Brief Title: Safety and Efficacy of ST-100 (Vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution in Subjects Diagnosed With Dry Eye Disease (DED)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: ORA, Inc. (Industry)
Collaborators: Stuart Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ST-100-002
Record Dates: First submitted 2023-12-07; First posted 2023-12-21 (Actual); Last update posted 2024-01-18 (Actual); Status verified 2024-01

CONDITIONS: Dry Eye Disease
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ST-100-002 (Experimental): ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Bilaterally twice daily for 7 weeks (49 days)
  Interventions: Drug: ST-100 (vezocolmitide)
- Vehicle Ophthalmic Solution (Placebo Comparator): Vehicle Ophthalmic Solution Bilaterally twice daily for 7 weeks (49 days)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: ST-100 (vezocolmitide) — ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml
  Arms: ST-100-002
Drug: Vehicle — Vehicle Ophthalmic Solution
  Arms: Vehicle Ophthalmic Solution

SUMMARY:
A Phase 3 Multi-Center, Randomized, Double Masked, Vehicle Controlled Study to Assess the Safety and Efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution in Subjects Diagnosed with Dry Eye Disease (DED)

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years of age;
2. Provide written informed consent;
3. Have a reported history of DED for at lease 6 months prior to Visit 1;
4. Have a history of use or desire to use eye drops for DED within 6 months of Visit 1;
5. Report a score of ≥ 2 on the Ora Calibra® Ocular Discomfort & 4-symptom questionnaire in at least one symptom pre-CAE® at Visits 1 and 2;
6. Have a Schirmer's Test score of ≤ 10 mm and ≥ 1 mm at Visits 1 and 2;
7. Have a conjunctival redness score ≥ 1 according to the Ora Calibra® Conjunctival Redness for Dry Eye Scale in at least one eye at pre-CAE® Visits 1 and 2;
8. Have a corneal fluorescein staining score of ≥ 2 in at least one region (e.g. inferior, superior, or central) pre-CAE® at Visits 1 and 2;
9. Have a sum corneal fluorescein staining score of ≥ 4, based on the sum of the inferior, superior, and central regions pre-CAE®, at Visits 1 and 2;
10. Have a total lissamine green conjunctival score of ≥ 2, based on the sum of the temporal and nasal regions pre-CAE® at Visits 1 and 2;
11. Demonstrates a response to the CAE® at Visits 1 and 2 as defined by:

    Having at least a ≥1 point increase in fluorescein staining in the inferior region in at least one eye following CAE® exposure Reporting an Ora Calibra® Ocular Discomfort Score ≥ 3 at 2 or more consecutive time points in at least one eye during CAE® exposure (if a subject has an ocular discomfort rating of 3 at a time = 0 for an eye, they must report an ocular discomfort rating of 4 for two consecutive measurements for that eye). Note: a subject cannot have an ocular discomfort score of 4 at time = 0);
12. Have at lease one single eye satisfy all criteria for 6, 7, 8, 9, 10 and 11 above.

Exclusion Criteria:

1. Have any clinically significant slit lap findings at Visit 1 that may include active blepharitis, meibomian gland dysfunction, lid margin inflammation, or active ocular allergies that require therapeutic treatment, and/or in the opinion of the investigator may interfere with study parameters;
2. Be diagnosed with an ongoing ocular infection (bacterial, viral, or fungal), or active ocular inflammation at Visit 1;
3. Have worn contact lenses within 7 days of Visit 1 or anticipate using contact lenses during the study;
4. Have used any eye drops within 2 hours of Visit 1;
5. Have previously had laser-assisted in situ keratomileusis (LASIK) surgery within the last 12 months;
6. Have used Restasis®, Xiidra®, or Cequa® ophthalmic solutions Tyrvaya® nasal spray, or Miebo® or Xdemvy® solution within 45 days of Visit 1;
7. Have any planned ocular and/or lid surgeries over the study period or any ocular surgery within the last 6 months;
8. Have used, are using or anticipate using permanent or temporary punctal plugs during the study within 90 days of Visit 1;
9. Be currently taking any topical ophthalmic prescription (including medications for glaucoma) or over-the-counter solutions, artificial tears, gels or scrubs, or using a moisture chamber and cannot discontinue these medications for the from Visit 1 until after Visit 8 of the trial (excluding medications allowed for the conduct of the study);
10. Be currently taking or have taken Omega-3 supplements within the last 3 months;
11. Be currently taking of have taken CHANTIX® (varenicline) tablets within 6 months prior to Visit 1 that is not on a stable dose. The dose cannot change during the conduct of the study;
12. Have corrected visual acuity (VA) greater than or equal to logarithm of the Minimum Angle of Resolution (logMAR) +0.7 as assessed by Early Treatment of Diabetic Retinopathy Study (ETDRS) scale in both eyes at Visit 1;
13. Be a woman who is pregnant, nursing, or planning a pregnancy during the study;
14. Be unwilling to submit a urine pregnancy test at Visit 1 and Visit 8 (or early termination visit) if of childbearing potential. Non-childbearing potential is defined as a woman who is permanently sterilized (hysterectomy, bilateral salpingectomy, bilateral oophorectomy at least 6 months prior to dosing), or is post-menopausal (where post-menopausal is defined as no menses for 12 months without an alternative medial cause);
15. Be a woman of childbearing potential who is not using an acceptable means of birth control; acceptable methods of contraception includes: hormonal - oral, implantable, injectable, or transdermal contraceptives for at least one month prior to first visit; Use two of the following effective methods of contraception: intrauterine device (IUD without local hormone release), diaphragm, cervical cap, and/or condoms; or surgical sterilization of partner (i.e., a female participant's male partner has undergone effective surgical sterilization such as vasectomy before the female participant entered the clinical trial) who has obtained documentation of absence of sperm in his ejaculate and is the sole sexual partner of the female participant during the clinical trial. For non-sexually active females, abstinence may be regarded as an adequate method of birth control; however, if the subject becomes sexually active during the study, she must agree to use adequate birth control as defined above for the remainder of the study;
16. Have a known allergy and/or sensitivity to the Study Drug or its components;
17. Have a condition or be in a situation that the investigator feels may put the subject at significant risk, may confound the study results, or may interfere significantly with the subject's participation in the study;
18. Be currently enrolled in an investigational drug or device study or have used an investigational drug or device within 30 days of Visit 1;
19. Be currently using any medication known to cause ocular drying that is not used on a stable dosing regimen for the least 30 dats prior to Visit 1;
20. Have a known history of meibomian gland procedures (e.g. LipiFlow, laser peripheral iridotomy (LPI), probing, etc.) within 6 months of study enrollment;
21. Be unable or unwilling to follow instructions, including participation in all study assessments and visits;
22. Has participated in any other clinical trials of ophthalmologic drugs for 30 days before or during participation in this Study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 175 (Estimated)
Dates: Start 2023-12-29 (Actual); Primary Completion 2024-06-30 (Estimated); Study Completion 2024-07-30 (Estimated)

PRIMARY OUTCOMES:
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle using Schirmer's test at day 29 | 29 Days
  Proportion of responders in Schirmer's test with ≥ 10mm improvement from baseline at Day 29

SECONDARY OUTCOMES:
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle for the treatment of the signs and symptoms of DED | 15 Days
  Ocular Discomfort scores change from baseline at day 15 as measured by Ora Calibra Ocular Discomfort Scale
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle for the treatment of the signs and symptoms of DED | 15 Days
  Pain Score change from baseline at Day 15
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle for the treatment of the signs and symptoms of DED | 4 days
  Blurred vision score change from baseline at day 4 as measured by OSDI
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle for the treatment of the signs and symptoms of DED | 15 days
  Proportion of responders in Schirmer's Test with ≥ 10mm improvement from baseline at day 15
Assess the safety and tolerability of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution | 49 days
  Visual Acuity
Assess the safety and tolerability of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution | 49 days
  Slit-lamp evaluation
Assess the safety and tolerability of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution | 49 days
  Adverse event monitoring
Assess the safety and tolerability of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution | 49 days
  Intraocular pressure
Assess the safety and tolerability of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution | 49 days
  Undilated fundoscopy

OTHER OUTCOMES:
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle using additional measures | 49 days
  Fluorescein staining (Ora Calibra scale) at Visits 3, 4, 5, 6, 7, and 8: regions: central, superior, inferior, temporal, nasal, corneal sum, conjunctival sum, and total eye score
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle using additional measures | 49 days
  Lissamine green staining (Ora Calibra scale) at Visits 3, 4, 5, 6, 7, and 8: regions: central, superior, inferior, temporal, nasal, corneal sum, conjunctival sum, and total eye score
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle using additional measures | 49 days
  Tear film break-up time at Visits 3, 4, 5, 6, 7, and 8
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle using additional measures | 49 days
  Conjunctival Redness at Visits 3, 4, 5, 6, 7, and 8
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle using additional measures | 49 Days
  Drop comfort assessment after randomization at Visit 2, 6, and 8
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle using additional measures | 49 Days
  Ocular Surface Disease Index (OSDI) at Visits 3, 4, 5, 6, 7, and 8
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle using additional measures | 49 days
  Ocular Discomfort Scale at Visits 3, 4, 5, 6, 7, and 8
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle using additional measures | 49 days
  Dry Eye Disease symptom questionnaire at Visits 3, 4, 5, 6, 7, and 8
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle using additional measures | 29 days
  Blink rate at Visits 6 and 7
Compare the efficacy of ST-100 (vezocolmitide) Ophthalmic Solution 60 μg/ml Ophthalmic Solution to vehicle using additional measures | 49 days
  Daily Dosing Diary

CONTACTS AND LOCATIONS:
Locations (1):
- Total Eye Care, PA, Memphis, Tennessee, United States

REFERENCES:
- [Result] Baratta RO, Schlumpf E, Buono BJD, DeLorey S, Calkins DJ. Corneal collagen as a potential therapeutic target in dry eye disease. Surv Ophthalmol. 2022 Jan-Feb;67(1):60-67. doi: 10.1016/j.survophthal.2021.04.006. Epub 2021 Apr 18. PMID 33882269
- [Result] Fiscella RG. Understanding dry eye disease: a managed care perspective. Am J Manag Care. 2011 Dec;17 Suppl 16:S432-9. PMID 22435675
- [Result] Hapach LA, VanderBurgh JA, Miller JP, Reinhart-King CA. Manipulation of in vitro collagen matrix architecture for scaffolds of improved physiological relevance. Phys Biol. 2015 Dec 21;12(6):061002. doi: 10.1088/1478-3975/12/6/061002. PMID 26689380
- [Result] Kivanany PB, Grose KC, Yonet-Tanyeri N, Manohar S, Sunkara Y, Lam KH, Schmidtke DW, Varner VD, Petroll WM. An In Vitro Model for Assessing Corneal Keratocyte Spreading and Migration on Aligned Fibrillar Collagen. J Funct Biomater. 2018 Sep 21;9(4):54. doi: 10.3390/jfb9040054. PMID 30248890
- [Result] Messmer EM. The pathophysiology, diagnosis, and treatment of dry eye disease. Dtsch Arztebl Int. 2015 Jan 30;112(5):71-81; quiz 82. doi: 10.3238/arztebl.2015.0071. PMID 25686388
- [Result] Ousler GW 3rd, Rimmer D, Smith LM, Abelson MB. Use of the Controlled Adverse Environment (CAE) in Clinical Research: A Review. Ophthalmol Ther. 2017 Dec;6(2):263-276. doi: 10.1007/s40123-017-0110-x. Epub 2017 Sep 27. PMID 28956287
- [Result] Shetty R, Deshpande K, Deshmukh R, Jayadev C, Shroff R. Bowman Break and Subbasal Nerve Plexus Changes in a Patient With Dry Eye Presenting With Chronic Ocular Pain and Vitamin D Deficiency. Cornea. 2016 May;35(5):688-91. doi: 10.1097/ICO.0000000000000785. PMID 26890669
- [Result] Wareham LK, Holden JM, Bossardet OL, Baratta RO, Del Buono BJ, Schlumpf E, Calkins DJ. Collagen mimetic peptide repair of the corneal nerve bed in a mouse model of dry eye disease. Front Neurosci. 2023 May 16;17:1148950. doi: 10.3389/fnins.2023.1148950. eCollection 2023. PMID 37260844